CLINICAL TRIAL: NCT02052154
Title: Multicenter Pilot Study Evaluating the Immunogenicity of an Innovative Pneumococcal Vaccination Strategy in Splenectomized Adults
Acronym: SPLENEVAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P120131; 2013-002631-19 (EudraCT Number)
Record Dates: First submitted 2014-01-20; First posted 2014-01-31 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Splenectomized Patients
Keywords: Pneumococcal infection; Splenectomized; vaccination
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prime-boost pneumococcal immunization (Experimental)
  Interventions: Biological: Prime-boost pneumococcal immunization

INTERVENTIONS:
Biological: Prime-boost pneumococcal immunization — 2 months between the 2 vaccines
  Other Names: Prevenar13® followed by Pneumo23®

SUMMARY:
Evaluate the immunogenicity of an innovative pneumococcal vaccination strategy in splenectomized adults comprising 1 dose of Prevenar13® conjugate vaccine (PCV) at M0 followed by 1 dose of Pneumo23® or Pneumovax® polysaccharide vaccine (PPSV) at M2. Duration of follow-up of 36 months.

The main endpoint will be the proportion of subjects responsive to 9 of the 13 serotypes common to the PCV and PPSV vaccines, selected because of their frequency in invasive infections in adults in France and their potentially reduced susceptibility to penicillin (serotypes 1, 3, 6A, 7F, 9V, 14, 19A, 19F, 23F).

DETAILED DESCRIPTION:
The splenectomized patient is more susceptible to infections because of the lack of specific response to the polysaccharide antigens that compose the capsules of certain bacteria. These very severe infections are known as Overwhelming Post Splenectomy Infections, or OPSI; they are characterized by very rapid onset with no prodrome and carry a high mortality rate. The annual incidence of OPSI is estimated at 0.23-0.42% with a lifetime risk of 5%. The role of pneumococcus in particular has been clearly established in these infections.

The most effective strategy to minimize the risk of pneumococcal infection is pneumococcal vaccination. Currently there are two types of vaccines available in France: polysaccharide and conjugate, both of which induce the production of anti-capsular IgG with both neutralizing and opsonic activity.

Since one of the consequences of asplenia is the absence of IgM production elicited by a polysaccharide challenge, due to an absence of splenic B cells, it is difficult to imagine that such patients would mount a satisfactory immune response to PPSV vaccination. And in fact, several studies have described the occurrence of pneumococcal OPSI in patients who were correctly vaccinated.

The study hypothesis is that a vaccination strategy combining PCV vaccine followed by PPSV vaccine will induce a good immune response in splenectomized patients, with good tolerability. All available data suggest that the optimum schedule consists of a primovaccination with one dose of PCV followed two months later by one dose of PPSV, in order to achieve a T-dependent memory response to the 13 serotypes common to the two vaccines.

The proposed endpoint is therefore to evaluate the immunogenicity and safety of a vaccination strategy comprising priming with one dose of Prevenar13® PCV vaccine (serotypes 4, 6B, 9V, 14, 18C, 19F, 23F, + 1, 3, 5, 6A, 7F, 19A) to induce a T cell memory response, followed by the classical administration of one dose of Pneumo23® or Pneumovax® vaccine (serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, 33F). Secondary endpoints will evaluate the safety of this strategy in terms of post-immunization local and systemic side effects, frequency of invasive pneumococcal infections, predictors of immunogenicity, and persistence of immunogenicity 30 months post-immunization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years
* Splenectomized since at least 2 weeks, with Howell-Jolly bodies on a blood smear and ultrasonographic confirmation
* No immunosppressived conditions : mainly trauma , idiopathic thrombocytopathic purpura or autoimmune hemolytic anemia, with no active treatment
* Available for 37 months of follow-up starting from the screening visit
* Contraception that the investigator judges effective for the first 2 months of the trial, with a negative pregnancy test
* Women not planning to become pregnant in the 6 months following inclusion (M0)
* Signed informed consent

Exclusion Criteria:

* Pregnancy or planned pregnancy in the 2 months following inclusion (M0)
* Pathology or conditions which modify immune response (excluding splenectomy) : HIV infection, immunosuppressive therapy ongoing or in 6 months before inclusion (M0), including corticosteroids > 10 mg daily, topic inhaled or dermic corticoid treatments are allowed, hematopoietic stem cell allo / autograft, primary immune deficiency, nephrotic syndrome, sickle cell disease, evolutive neoplasia
* History of anaphylactic reaction following vaccination
* Known allergy to any of the ingredients of the vaccines: aluminium phosphate, phenol, Corynebacterium diphtheriae CRM-197 protein
* Previous vaccination with 7-valent or 13-valent pneumococcal conjugate vaccine (in the 5 last years)
* Previous vaccination with the pneumococcal polysaccharidic vaccine in the 3 years before inclusion (M0)
* Other vaccination in the month before inclusion (M0)
* Polyvalent immunoglobulin infusion in the 3 months before inclusion (M0) or during the planned duration of the study
* Anticoagulant treatment current or stopped less than 7 days before inclusion (M0); or clotting disorder contra-indicating intramuscular injection
* Participation to an other vaccine study in the 28 days before inclusion till the end of study
* Not covered by national health insurance (beneficiary or assignee)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects responsive to 9 of the 13 serotypes common (serotypes 1, 3, 6A, 7F, 9V, 14, 19A, 19F, 23F). | M3
  According to currently accepted international guidelines, a subject is considered to be responsive to a given serotype if one month after PPSV vaccination (at M3) the specific IgG titer is ≥ 1 μg/mL by ELISA and the opsonophagocytosis assay (OPA) threshold response is ≥ at LLOQ (Lower limit of quantification)

SECONDARY OUTCOMES:
IgG dosage | one month
  Immunologic Response after one injection PnCj (Specific IgG ≥1 µg/ml)
ELISA dosages | 4 months after PPSV vaccine
  Evaluation of persistent responses 4 months after PPSV vaccine
ELISA dosages | 10 months after PPSV vaccine
  Evaluation of persistent responses 10 months after PPSV vaccine
ELISA dosages | 34 months after PPSV vaccine
  Evaluation of persistent responses 34 months after PPSV vaccine
Identification of predictive factors for immunogenicity | M0 to M36
  Identification of predictive factors for immunogenicity: age, gender, indication for splenectomy, time since splenectomy, time since previous vaccination with polysaccharide vaccine, number of PPSV vaccinations previously received
Percentage of patients presenting local or systemic reactions post-immunization | M0 to M36
  Estimate the clinical and biological tolerance of the vaccinal strategy
Evaluation of severe infectious episode | M0 to M36
  the evaluation of severe infectious episode are assessed with microbiological documentation (with serotype if Streptococcus pneumoniae), site of infection, occurrence under antibiotic prophylaxis or not.
  this will allow to list and characterize the serotype involved during possible episodes of invasive infections in pneumocoque
OPA dosages | 4 months after PPSV vaccine
  Evaluation of persistent responses 4 months after PPSV vaccine
OPA dosages | 10 months after PPSV vaccine
  Evaluation of persistent responses 10 months after PPSV vaccine
OPA dosages | 34 months after PPSV vaccine
  Evaluation of persistent responses 34 months after PPSV vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Hélène COIGNARD-BIEHLER, MD, Principal Investigator — Service des Maladies Infectieuses et Tropicales, Hôpital Necker-Enfants Malades, APHP; Olivier LORTHOLARY, MD, PhD, Study Director — Service des Maladies Infectieuses et Tropicales, Hôpital Necker-Enfants Malades, APHP; Odile LAUNAY, MD, PhD, Study Director — CIC Vaccinologie Cochin-Pasteur (CIC BT505) - Hôpital Cochin; Marc MICHEL, MD, PhD, Study Director — Service de médecine interne, Hôpital Henri Mondor; Frédéric BATTEUX, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Claude-Agnès REYNAUD, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Pierre BUFFET, MD, PhD, Study Chair — INTS
Locations (1):
- Service des Maladies Infectieuses et Tropicales - Centre d'Infectiologie Necker-Pasteur, IHU Imagine - Hôpital Necker-Enfants, Paris, France